CLINICAL TRIAL: NCT06514690
Title: Postoperative Memories and Optimal Level of Sedation for Tracheal Intubation Using Fiberoptic Bronchoscopy/Vidolaryngoscopy in Patients With Anticipated Difficult Airway Undergoing Surgery
Brief Title: Postoperative Memories and Level of Sedation for Tracheal Intubation Using Fiberoptic Bronchoscopy/Videolaryngoscopy
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: EOM(AG)014/2023(6107)
Record Dates: First submitted 2023-04-29; First posted 2024-07-23 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Difficult Airway; Postoperative Memories; Tracheal Intubation
Keywords: postoperative memories; tracheal intubation; difficult airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients intubated by fiberoptic bronchoscope: Fiberoptic bronchoscopy involves the introduction of a flexible tube (bronchoscope) through the nose that has a light and a video camera at its tip. It allows directing the orotracheal tube into the airway.
  Interventions: Other: Sedation
- Patients intubated by videolaryngoscopy: The videolaryngoscopy allows tracheal intubation by introducing a laryngoscope and visualizing the glottis on an external display.
  Interventions: Other: Sedation

INTERVENTIONS:
Other: Sedation — Different degrees of intravenous sedation according to the Ramsay scale

SUMMARY:
Antecedentes In patients with expected difficult airways undergoing surgery, tracheal intubation must be performed with a fiberoptic bronchoscope or video laryngoscope while keeping the patient awake and under the effects of anesthetic sedation.

Objective: To determine and compare the existence of postoperative memories of the patients and the different levels of sedation (Ramsay scale) obtained during the intubation procedure.

Methods Prospective observational study that includes 100 patients older than 18 years who are going to undergo surgery, who need fiberoptic bronchoscopy/videolaryngoscopy for tracheal intubation due to the planned difficult airway and intravenous sedation. Patients with an unexpected difficult airway, under 18 years of age and/or with cognitive impairment will be excluded. After checking the tracheal intubation, the general anesthesia indicated for each patient will be used.

Twenty-four hours after tracheal extubation, the patient will be questioned about the pain presented during the fiberoptic bronchoscopic/videolaryngoscopic procedure and postoperative memories based on a modified Brice questionnaire. At 30 days after surgery, the postoperative memories of the patients will be evaluated again by telephone interview.

DETAILED DESCRIPTION:
Background In patients with expected difficult airways undergoing surgery, tracheal intubation must be performed with a fiberoptic bronchoscope or video laryngoscope while keeping the patient awake and under the effects of anesthetic sedation. The intravenous sedation has the advantages of relieving anxiety, providing maximum comfort to the patient, facilitating examination, and producing amnesia of the episode. As an inconvenience, it can produce a depression of the respiratory system, fearsome in patients with expected difficult airway. Given the fear of the appearance of respiratory depression in these patients, the levels of sedation achieved are usually not very deep, and there may be pain and the presence of unpleasant postoperative memories in relation to the intubation technique using bronchoscopy/videolaryngoscopy.

Main objective: To determine and compare the existence of postoperative memories of patients who need conscious tracheal intubation, but under the effects of sedation, due to the planned difficult airway, depending on whether intubation was performed with a fiberoptic bronchoscope or video laryngoscope.

Secondary objective: To determine if there is a relationship between the appearance of postoperative memories and the different levels of sedation (Ramsay scale) obtained during the intubation procedure.

Other objectives: To determine if the duration of tracheal intubation time influences the incidence of postoperative memories. Determine the incidence of respiratory depression (SpO2 <90%) during the tracheal intubation procedure. Pain presented by patients during the procedure.

Methods Prospective observational study

Inclusion criteria:

* Patients older than 18 years
* Patients with predicted difficult airway who need surgery
* Patients undergoing tracheal intubation using fiberoptic bronchoscopy/videolaryngoscopy

Exclusion criteria:

* Patients <18 years.
* Patients without expected difficult airway
* Patients with cognitive impairment, Informed consent for anesthesia will specify the need for fiberoptic bronchoscopy/videolaryngoscopy for tracheal intubation and will require the patient's written authorization to participate in this study.

Before performing fiberoptic bronchoscopy/videolaryngoscopy, the patient will be monitored (blood pressure, ECG, SpO2) and O2 will be administered to try to maintain SpO2 levels above 90%. Next, we will proceed to intravenous sedation. After checking the tracheal intubation, the general anesthesia indicated for each patient will be used.

The level of sedation obtained during the tracheal intubation procedure can be any of those classified on the Ramsay scale, at the discretion of the anesthesiologist.

For each study group (fibrebronchoscope-videolaryngoscope) the following will be recorded: the demographic characteristics of the patients; the type of surgery and its duration; duration of fiberoptic bronchoscopy/videolaryngoscopy; intravenous sedation drugs administered and their doses; nasal (instillation, spray), pharyngeal (spray) and/or vocal cord (instillation) administration of lidocaine; the existence of respiratory depression (lower peripheral oxygen saturation (SpO2) level); the highest and lowest systolic blood pressure (SBP) and heart rate (HR) values; the lowest bispectral index (BIS) value; and the time that the patient remains intubated after surgery.

Twenty-four hours after tracheal extubation, the patient will be questioned about the pain presented during the fiberoptic bronchoscopic/videolaryngoscopic procedure and postoperative memories based on a modified Brice questionnaire. At 30 days after surgery, the postoperative memories of the patients will be evaluated again by telephone interview.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients undergoing surgery
* Patients with predicted difficult airway

Exclusion Criteria:

* Patients under 18 years of age
* Patients without cognitive disorders

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years undergoing surgery, who need fiberoptic bronchoscopy/videolaryngoscopy for tracheal intubation due to the planned difficult airway and intravenous sedation.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2025-04-29 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
Incidence of postperative memories | 24 hours after tracheal extubation and 30 days after
  * Determine and compare, between study groups, the existence of postoperative memories according to Brice's questionnaire, in patients who need conscious tracheal intubation, under the effects of intravenous sedation.
  * Determine and compare, between study groups, postoperative memories for each sedation level of the Ramsay scale.

SECONDARY OUTCOMES:
Determine other adverse effects: | during fiberoptic bronchoscopy/videolaryngoscopy procedure
  Record patients who present respiratory depression (SpO2 <90%), discomfort (cough and movements)

CONTACTS AND LOCATIONS:
Locations (1):
- Susana González Suárez, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No